CLINICAL TRIAL: NCT06768411
Title: The Dosage Exploration Study of PEG-rhGH for Treating Short Stature in Prepubertal and Pubertal Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAHoWMU-CR2024-06-223
Record Dates: First submitted 2024-12-24; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Short Stature
MeSH Terms: conditions — Dwarfism | interventions — polyethylene glycol-recombinant human growth hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- prepubertal children of short stature (Other): prepubertal children of short stature with different Initial doses of PEG-rhGH
  Interventions: Drug: PEG-rhGH
- pubertal children of short stature (Other): pubertal children of short stature with different Initial doses of PEG-rhGH with or without GnRHa treatment
  Interventions: Drug: PEG-rhGH; Drug: GnRHa

INTERVENTIONS:
Drug: PEG-rhGH — 1= 0.2mg/kg/week Initial doses of PEG-rhGH 2=0.22mg/kg/week Initial doses of PEG-rhGH
  Other Names: 1; 2
Drug: GnRHa — 1. pubertal children of short stature without GnRHa treatment
  2. pubertal children of short stature with GnRHa treatment
  Arms: pubertal children of short stature

SUMMARY:
This study is dedicated to addressing the lack of research on the most effective dosage of long-acting growth hormone for children with short stature. By employing clinical trial design, we are committed to investigating the therapeutic benefits and safety profiles associated with varying doses of long-acting growth hormone. Our ultimate goal is to offer clinicians more precise treatment guidance and assist patients in attaining optimal growth and developmental outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with short stature or a genetic target height below 2 standard deviations;
2. Individuals who are pre-pubertal (Tanner stage I) and pubertal (Tanner stages II-IV).
3. Legal guardians consenting to participate in the study and signing informed consent forms.

Exclusion Criteria:

1. Known or suspected hypersensitivity reactions to the investigational product or related products;
2. Presence of severe systemic diseases;
3. Patients with malignant tumors;
4. Participation in any other clinical trial and receipt of drug or non-drug interventions within the 3 months prior to screening;
5. Patients unable to adhere to follow-up or receive treatment as scheduled;
6. Other circumstances in which the investigator deems the patient unsuitable for inclusion in this clinical trial.

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
height growth rate | 2 years
  Measure the height and observe how many centimeters it grows each month

SECONDARY OUTCOMES:
Sexual development status | two years
  Evaluate Tanner staging, The Tanner Staging, also known as Sexual Maturity Rating (SMR), is a classification system that healthcare providers use to document and track the development of secondary sex characteristics of children during puberty. It's a tool that outlines the stages of puberty for children and when they're likely to occur.
IGF-1 | two years
  IGF-1, known as insulin-like growth factor, is utilized to evaluate the efficacy of growth hormone therapy. By measuring IGF-1 levels, doctors can determine the effectiveness of the treatment and whether the patient's growth falls within the normal range

OTHER OUTCOMES:
bone age | 2 years
  Bone age assessment